CLINICAL TRIAL: NCT04456868
Title: Neurophysiological Markers in the Depressive Episode Characterized by Anhedonic Drug Resistance: Evaluation of Motor Skills and P300 Wave
Acronym: PHYDDOPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to include additional patients in the arms with depression
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/0426/HP
Record Dates: First submitted 2020-03-16; First posted 2020-07-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bipolar Anhedonic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers (Active Comparator): Healthy volunteers at least 18 years old and without a history of psychiatric or neurological disorders
  Interventions: Behavioral: Electroencephalogram; Behavioral: walking test; Behavioral: Quality of life questionnaire
- Anhedonic drug-resistant bipolar depression patient (Experimental): Adult patients at least 18 years old with drug-resistant bipolar depression of the anhedonic type
  Interventions: Behavioral: Electroencephalogram; Behavioral: walking test; Behavioral: Quality of life questionnaire; Procedure: Position emission tomography
- Non-anhedonic drug-resistant bipolar depression Pat (Active Comparator): Adult patients at least 18 years old with drug-resistant bipolar depression of the non-anhedonic type
  Interventions: Behavioral: Electroencephalogram; Behavioral: walking test; Behavioral: Quality of life questionnaire; Procedure: Position emission tomography
- Mild to moderate Parkinson's disease patient (Active Comparator): Adult patients at least 18 years of age with mild to moderate Parkinson's disease
  Interventions: Behavioral: Electroencephalogram; Behavioral: walking test; Behavioral: Quality of life questionnaire; Procedure: Position emission tomography

INTERVENTIONS:
Behavioral: Electroencephalogram — Electroencephalogram will be done for P300 wave assessment
Behavioral: walking test — 8-Meter walking test will be done for gait parameter assessment
Behavioral: Quality of life questionnaire — Starkstein Apathy Scale, DSM-5 criteria, Montgomery-Åsberg Depression Rating Scale, Perseverative Thinking Questionnaire, classification of Hoehn & Yahr
Procedure: Position emission tomography — Position emission tomography will be done for
  Arms: Anhedonic drug-resistant bipolar depression patient; Mild to moderate Parkinson's disease patient; Non-anhedonic drug-resistant bipolar depression Pat

SUMMARY:
Depression is currently the leading cause of disability and suicide death worldwide. Several studies, however, have shown that a significant proportion of patients do not respond to standard antidepressants, especially since their symptomatology is dominated by anhedonia or psychomotor retardation reflecting central dopaminergic dysfunction. In order to improve the efficiency and speed of the antidepressant response, it seems essential to highlight this dopaminergic dysfunction, by defining a P300 wave profile specific to the subtype of depressed patients with anhedonic phenotype to whom personalized treatment targeting dopaminergic transmission could in the future be proposed earlier. The investigators therefore wish to highlight an increase in the latency time of P300 and a modification of motor skills (of the walking cycle and of the movement of the hands), without modification of the dopaminergic transmission measured by PETScan, specific to the sub-type of depressive patients, resistant to at least 2 antidepressants of different classes with an anhedonia score> 5/14 on the SHAPS scale. The increased latency of P300 could then be used in the future as a predictive biomarker of resistance to conventional antidepressant treatments specific to this population of anhedonic depressed patients

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:
* Person who is ≥ 18 years old and ≤ 70 years old
* Subject without neurological history
* Subject without psychiatric history in the semi-structured interview Mini International Neuropsychiatric Interview (MINI).
* Subject having read and understood the newsletter and signed the consent form
* Subject affiliated to a social security scheme.
* Subject capable of understanding spoken and written French.
* Woman of reproductive age with effective contraception as defined by the WHO, for at least three months or postmenopausal.

Patients with drug-resistant bipolar anhedonic depression:

* Patient whose age is ≥ 18 years and ≤ 70 years.
* Patient with depression meeting DSM-5 criteria (Appendix 4) evolving in the context of bipolar disorder.
* Patient with a resistance level greater than or equal to 1 according to the Pacchiarotti classification.
* Patient with an SHAPS anhedonia score greater than 5/14.
* Patient with no other psychiatric pathology in the semi-structured interview Mini International Neuropsychiatric Interview (MINI).
* Stable lithium treatment in the 7 days preceding the inclusion visit.
* Patient who has not received treatment with electroconvulsive therapy in the 2 months preceding the inclusion visit.
* Patient having a normal neurological examination.
* Patient who has read and understood the information letter and signed the consent form.
* Patient affiliated to a social security scheme.
* Patient able to understand spoken and written French.
* Woman of reproductive age with effective contraception as defined by the WHO, for at least three months or postmenopausal.Patient dont l'âge est ≥ 18 ans et ≤ 70 ans.

Patients with drug-resistant bipolar depression of the non-anhedonic type:

* Patient whose age is ≥ 18 years and ≤ 70 years.
* Presence of a depression meeting the criteria of DSM-5 (Annex 4) evolving in the context of bipolar disorder.
* Patient with a resistance level greater than or equal to 1 according to the Pacchiarotti classification.
* Patient with SHAPS anhedonia score less than or equal to 3/14.
* Absence of another psychiatric pathology in the semi-structured interview Mini International Neuropsychiatric Interview (MINI).
* Stable lithium treatment in the 7 days preceding the inclusion visit.
* Patient who has not received treatment with electroconvulsive therapy in the 2 months preceding the inclusion visit.
* Patient having a normal neurological examination.
* Patient who has read and understood the information letter and signed the consent form.
* Patient affiliated to a social security scheme.
* Patient able to understand spoken and written French.
* Woman of reproductive age with effective contraception as defined by the WHO, for at least three months.

Patients with Parkinson's disease :

* Patient whose age is ≥ 18 years and ≤ 70 years.
* Patient with idiopathic Parkinson's disease as defined by the diagnostic criteria of the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) (Annex 8).
* Patient with Parkinson's disease stage less than 3 (mild or moderate severity) according to the classification of Hoehn & Yahr (Annex 7).
* Patient treated with L-DOPA associated with a dopa-decarboxylase inhibitor (DDC) and who has not changed antiparkinsonian treatment for at least 1 month before the inclusion visit.
* Patient with no neurological disorders other than those induced by Parkinson's disease.
* Patient without depression defined by a score less than or equal to 8 on the Montgomery-Åsberg Depression Rating Scale (MADRS) (Annex 10).
* Patient with no psychiatric pathology at the semi-structured interview Mini International Neuropsychiatric Interview (MINI) (Annex 9).
* Patient who has read and understood the information letter and signed the consent form.
* Patient affiliated to a social security scheme.
* Patient able to understand spoken and written French.
* Woman of childbearing age with effective contraception as defined by the WHO, for at least three months.

Exclusion Criteria:

* Healthy volunteers:
* Person with a psychiatric disorder in the semi-structured interview Mini International Neuropsychiatric Interview (MINI) (Annex 9).
* Person deprived of their liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship.
* Subjects with poor understanding of spoken or written French
* Existence of a neurological, rheumatological, orthopedic or psychiatric history, presence of a severe progressive pathology which can modify brain activity or gait parameters.
* Woman of childbearing age not taking effective contraception according to the WHO definition (estrogen-progestogens or intrauterine device or tubal ligation), pregnant (positive urine pregnancy test) or breastfeeding.
* Taking unauthorized treatment during the study and:

  * In the 7 days preceding inclusion for dopamine agonists, MAOIs, antiepileptics, antidepressants, benzodiazepines and L-DOPA combined with a dopa decarboxylase (DDC) or catechol-O-methyl transferase inhibitor (COMT).
  * In the 28 days preceding inclusion for amphetamines, antivirals, antiemetics.
  * In the 2 months preceding inclusion for electroconvulsive therapy
  * In the 6 months prior to inclusion for antipsychotics.
* Dependence on a substance other than nicotine.

Patients with drug-resistant bipolar anhedonic depression:

* Patient with depression with psychotic characteristics.
* Patient deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship.
* Subjects with poor understanding of spoken or written French
* Patient with SHAPS anhedonia score less than or equal to 5/14 (Annex 2).
* Patient with a neurological, rheumatological, orthopedic or psychiatric history, presence of a severe progressive pathology which can modify brain activity or gait parameters.
* Woman of childbearing age not taking effective contraception according to the WHO definition (estrogen-progestogens or intrauterine device or tubal ligation), pregnant (positive urine pregnancy test) or breastfeeding.
* Subject with a history of allergy or hypersensitivity to the active substance in DOPACIS (18Fluorodopa) or to any of its excipients.
* Taking unauthorized treatment during the study and:

  * In the 7 days preceding inclusion for dopamine agonists, MAOIs, antiepileptics, antidepressants, benzodiazepines and L-DOPA combined with a dopa decarboxylase (DDC) or catechol-O-methyl transferase inhibitor (COMT).
  * In the 28 days preceding inclusion for amphetamines, antivirals, antiemetics.
  * In the 2 months preceding inclusion for electroconvulsive therapy
  * In the 6 months prior to inclusion for antipsychotics.
* Dependence on a substance other than nicotine.

Patients with drug-resistant bipolar depression of the non-anhedonic type:

* Pa Patient with depression with psychotic characteristics.
* Patient deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship.
* Subjects with poor understanding of spoken or written French
* Patient with SHAPS anhedonia score less than or equal to 5/14 (Annex 2).
* Patient with a neurological, rheumatological, orthopedic or psychiatric history, presence of a severe progressive pathology which can modify brain activity or gait parameters.
* Woman of childbearing age not taking effective contraception according to the WHO definition (estrogen-progestogens or intrauterine device or tubal ligation), pregnant (positive urine pregnancy test) or breastfeeding.
* Subject with a history of allergy or hypersensitivity to the active substance in DOPACIS (18Fluorodopa) or to any of its excipients.
* Taking unauthorized treatment during the study and:

  * In the 7 days preceding inclusion for dopamine agonists, MAOIs, antiepileptics, antidepressants, benzodiazepines and L-DOPA combined with a dopa decarboxylase (DDC) or catechol-O-methyl transferase inhibitor (COMT).
  * In the 28 days preceding inclusion for amphetamines, antivirals, antiemetics.
  * In the 2 months preceding inclusion for electroconvulsive therapy
  * In the 6 months prior to inclusion for antipsychotics.
* Dependence on a substance other than nicotine.

Patients with Parkinson's disease:

* Patient with depression.
* Patient deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-tutorship or curatorship.
* Subjects with poor understanding of spoken or written French
* Severe form of Parkinson's disease with a Hoehn and Yhar upper or equal 4 (Annex 7).
* Patient with other neurological, rheumatological, orthopedic or psychiatric history, presence of a severe progressive pathology which can modify brain activity or gait parameters.
* Woman of childbearing age not taking effective contraception according to the WHO definition (estrogen-progestogens or intrauterine device or tubal ligation), pregnant (positive urine pregnancy test) or breastfeeding.
* Subject with a history of allergy or hypersensitivity to the active substance in DOPACIS (18Fluorodopa) or to any of its excipients.
* Taking unauthorized treatment during the study and:

  * In the 7 days preceding inclusion for dopamine agonists, MAOIs, antiepileptics, antidepressants, benzodiazepines and L-DOPA combined with a dopa decarboxylase (DDC) or catechol-O-methyl transferase inhibitor (COMT).
  * In the 28 days preceding inclusion for amphetamines, antivirals, antiemetics.
  * In the 2 months preceding inclusion for electroconvulsive therapy
  * In the 6 months prior to inclusion for antipsychotics.
* Dependence on a substance other than nicotine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Difference between latency of P300 wave during encephalogram | 1 hour after inclusion

SECONDARY OUTCOMES:
Difference in walking speed during an 8 meter-walk test between the group of patients with bipolar drug-resistant depression of the anhedonic type and the other groups of subjects | 2 hours after inclusion
Stride length variation during an 8 meter-walk test between the group of patients with bipolar drug-resistant depression of the anhedonic type and the other groups of subjects | 2 hours after inclusion
Difference in presynaptic fixation of 18-Fluorodopa during positron emission tomography between the group of patients with drug-resistant bipolar depression of the anhedonic type and the other groups of patients | 4 hours after inclusion
Difference in the apathy assessment score performed by the Starkstein Apathy Scale (SAS) between the group of patients with drug-resistant bipolar depression of the anhedonic type and the other groups of subjects | 30 minutes after inclusion
  Starkstein Apathy Scale (SAS) is scored from 0 to 42 42 = maximum severity of apathy ; Score <14 define a absence apathy Score ≥14 define the presence of a clinically significant apathy
Difference in frequency of melancholic characteristics meeting the criteria of DSM-5 between the group of patients with drug-resistant bipolar depression of the anhedonic type and the other groups of subjects | 30 minutes after inclusion
  melancholic characteristics of DSM-5 has 8 items (2 A catory and 6 B category) Presence of melancholic characteristics is defined by a presence of at least one item from A category and the presence of at least 3 items from B category Absence of melancholic characteristics is defined by no item from A category and less than 3 items from B category
Difference in the Montgomery-Åsberg Depression Rating Scale (MADRS) assessment score for EDC severity between the group of patients with bipolar drug-resistant depression of the anhedonic type and the other groups of subjects | 30 minutes after inclusion
  Montgomery-Åsberg Depression Rating Scale (MADRS) 10 items scored from 0 to 6 (6 correspond to maximal severity of the item). The score varies from 0 to 60 (60 = maximal severity of intensity of depression).
  Total score ≥ 8/60 defines a clinically significant intensity of depression. Total score > 30/60 defines a major intensity of depression
Difference in the score for evaluation of repetitive negative thinking by the Perseverative Thinking Questionnaire (PTQ) between the group of patients with bipolar drug-resistant | 30 minutes after inclusion
  the Perseverative Thinking Questionnaire (PTQ) has 15 items scored from 0 (never) to 5 (almost always = maximum severity of the dimension evaluated by the item). The score varies from 0 (absence of repetitive negative thinking) to 60 (maximum severity of the intensity of repetitive negative thinking)
Difference in the score for the evaluation of parkinsonian symptoms (classification of Hoehn & Yahr) between the group of patients with bipolar drug-resistant depression of the anhedonic type and the other groups of patients | 30 minutes after inclusion
  The score varies from 0 (no sign) to 5 (worse disability)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure WELTER, Pr, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Rouen University Hospital, Rouen
  - CHSR du Rouvray, Saint-Étienne-du-Rouvray

IPD SHARING:
Plan to Share IPD: No